CLINICAL TRIAL: NCT05957146
Title: Kinetics of Extracellular Vesicles in Hemodialysis
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dianet Dialysis Centers (Other)
Responsible Party: Principal Investigator, Muriel P.C. Grooteman, Principal investigator, MD PhD, Amsterdam UMC, location VUmc
Other Study IDs: NL84115.018.23
Record Dates: First submitted 2023-07-04; First posted 2023-07-24 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: End-stage Kidney Disease
Keywords: Hemodialysis; Extracellular vesicles; Bio-incompatibility; Tissue injury
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic hemodialysis patients: Adult patients treated with routine hemodialysis 3x/week during at least 3 months
  Interventions: Device: Routine hemodialysis

INTERVENTIONS:
Device: Routine hemodialysis — * Dialyzers: Cordiax FX80 dialyzers; membrane material HelixonePlus (polysulfone); (Fresenius Medical Care Bad Homburg, Germany)
  * Dialysis machines: Baxter Gambro AK 98 (Gambro Lundia AB, Lund, Sweden; part of Baxter Healthcare Corporation)
  * Needles for vascular access: Nipro SafeTouch dialysis cath 1.6x25 mm (16G) or 1.9x25 mm (15G); or Nipro SafeTouch Tulip needles (15G; all Nipro Medical Europe Mechelen, Belgium)
  * Ultrapure dialysis fluids (less than 0.1 colony forming units/ml, less than 0.03 endotoxin units/ml) will be mixed with AC-F 219/1 or 213/4 liquid acid concentrates and BiBag dry bicarbonate concentrate. Hence, the electrolyte composition of the dialysis fluid will be: Na 138-142 mmol/L; K 2.0-3.0 mmol/L; HCO3 26-35 mmol/L; Ca 1.25-1.50 mmol/L; Mg 0.5 mmol/L; Cl 108.5-109 mmol/L; glucose 5.6 mmol/L; acetate 3 mmol/L. Dialysate flow rate will be 500 mL/min.
  * Anticoagulation: nadroparin.

SUMMARY:
The aim of this observational study is to gain insight into the kinetics of extracellular vesicles (EVs), derived from both in- (i.e. bio-incompatibility) and outside (tissue-injury) the extracorporeal circuit (ECC), during standard hemodialysis (HD) in adult prevalent end-stage kidney disease (ESKD) patients treated with HD.

During a single HD session, blood samples for EV-assessment will be taken at several time points and at different sampling sites in the extracorporeal circuit (sampling point 1: before the rollerpump, arterial line; sampling point 2: after the rollerpump and before the dialyzer, sampling point 3: after the dialyzer, efferent line).

DETAILED DESCRIPTION:
Hemodialysis (HD) is a lifesaving treatment for ESKD patients. Yet, apart from beneficial effects, HD has adverse consequences, which, apart from rapid osmolality and electrolyte shifts, results from the bio-incompatibility (BI) of the extra-corporeal circuit (ECC) and intradialytic hypotension (IDH) as well. While BI arises within the ECC due to the contact between circulating blood cells and the foreign materials of the lines and dialyzer, IDH-induced tissue injury (TI) originates within the body of the patients. Activated cells can be detected by upregulation of cell surface markers and release of degradation products. Substances which are smaller than the pores of dialyzer-membranes may pass this barrier and, thus, become undetectable in blood.

Various cell types shed small particles upon activation an/or injury, so called extracellular vesicles (EVs). These EVs, which are shed by various cell types upon activation and/or injury, contain various proteins and are too large to travers dialyzer membranes. Their assessment requires strict and standardized collection and handling of blood samples. In previous HD research, both pre-analytical circumstances and analytic methods were insufficiently standardized, precluding solid conclusions. Both the contact between circulating blood cells and the ECC, and recurrent IDH, predispose to micro-inflammation and cell activation, which are related to morbidity and mortality. Hence, when analysed properly, the measuring of EVs might be a valuable tool to assess dialysis-induced adverse side-effects, not only in the dialyzer but also in the body, which, when occurring repeatedly, may influence survival.

In a recent study, we found an increase in EVs during treatment with different dialysis modalities. However, EVs were only assessed before and after dialysis. Hence, in the present study, we aim to assess the kinetics of EVs in routine HD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Stable clinical situation: free of infection, no recent admission
* HD >3 months
* Haemoglobin level >6,2 mmol/L
* Residual diuresis <200mL/24h
* Willing and able to give written informed consent.

Exclusion Criteria:

* Active infection, malignancy, auto-immune disease, or treatment with immunosuppressive medication.
* Allergy to polysulfone dialysers
* Life expectancy <3 months due to non-renal disease
* Access recirculation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients treated with chronic intermittent hemodialysis (3x per week during 4 hours) during at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Intradialytic change in the concentration of extracellular vesicles from specific cell types | 4 hours (=one dialysis treatment); assessed at the following time points: 0 minutes (start of dialysis), 30 min, 60 min, 120 min, 180 min, 235 minutes
  Blood cell-derived EVs: platelets: CD61+, activated platelets: CD61+/CD62p+; erythrocytes: CD235a+; leukocytes CD45+; and endothelium-derived EVs: CD144+, activated endothelium CD62e+; myocardium and endothelium-derived: Connexin-43+ will be measured at different sampling sites (sampling point 1: before the roller pump, arterial line; sampling point 2: after the rollerpump and before the dialyzer, sampling point 3: after the dialyzer, efferent line).

SECONDARY OUTCOMES:
Intradialytic blood pressure | 4 hours (=one dialysis treatment); measured 4x/hour
  Change in systolic and diastolic blood pressure (mmHg) during dialysis
Hematocrit (Ht) | 4 hours (=one dialysis treatment); measured three times (at the start (0 minutes), half way (120 minutes) and at the end (240 minutes))
  the volume percentage of red blood cells (RBCs) in blood
High sensitive CRP (hsCRP) | 4 hours (=one dialysis treatment); measured once at the start of dialysis (0 minutes)
  Marker of inflammation
White blood cell (WBC) count | 4 hours (=one dialysis treatment); measured once at the start of dialysis (0 minutes)
  Total white blood cell count and differential count
Platelet count | 4 hours (=one dialysis treatment); measured once at the start of dialysis (0 minutes)
  Number of platelets in blood

CONTACTS AND LOCATIONS:
Overall Officials: Muriel PC Grooteman, MD PhD, Principal Investigator — VUmc
Locations (1):
- Dianet Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No